CLINICAL TRIAL: NCT07200713
Title: A Randomized Controlled Evaluation of Sensory Motor Arousal Regulation Treatment (SMART) for Youth With Developmental Trauma and Self-regulation Difficulties
Brief Title: Effect Study of SMART Treatment for Youth
Acronym: UTVID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 881408
Record Dates: First submitted 2025-09-10; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Stress Disorders, Traumatic; Psychological Trauma; Sexual Trauma; Stress Disorders, Post-Traumatic; Mental Disorders
Keywords: Randomized controlled trial; Developmental trauma disorder; self-regulation difficulties; trauma treatment; Sensory motor arousal regulation treatment (SMART); Children; Youth; Outpatient treatment; Treatment as usual
MeSH Terms: conditions — Stress Disorders, Traumatic; Psychological Trauma; Sexual Trauma; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: At each of four study sites, the study uses blocked randomization with alternating block sizes of 4 and 6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory motor arousal regulation treatment (SMART) (Experimental): Treatment using SMART rooms and associated SMART techniques
  Interventions: Other: Sensory motor arousal regulation treatment (SMART)
- Treatment as usual (TAU) (Active Comparator): Best practice ordinary treatment without using SMART approaches
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Other: Treatment as usual (TAU) — Best practice ordinary psychological treatment
  Arms: Treatment as usual (TAU)
Other: Sensory motor arousal regulation treatment (SMART) — Psychological treatment using SMART room and associated techniques
  Arms: Sensory motor arousal regulation treatment (SMART)

SUMMARY:
The goal of this clinical trial is to learn if Sensory motor arousal regulation treatment (SMART) works better than treatment as usual (TAU) to treat youth 7-17 years with complex trauma histories and self-regulation difficulties. The study also will investigate which patients will benefit more from SMART (treatment effect heterogeneity) and whether therapeutic alliance mediates effect. The main hypotheses the trial aims to answer are:

1. Main effects: The SMART model approach will be more effective than ordinary treatment (control condition), in terms of improvement from therapy starts to 6 and 12 months follow up, for:

   1. Regulatory capacities of emotions and bodily states, attention and behavior, and self and social relations
   2. Trauma symptoms of re-experiencing, avoidance/ numbness and hyperarousal and sense of threat (core PTSD symptoms) and disturbances in self-organization (affect, self-concept; relations - core complex PTSD symptoms)
   3. Internalizing symptoms (somatic complaints, anxiety symptoms and depression symptom severity) and Externalizing symptoms (conduct problems, aggression, inattention, and social problem severity)
   4. Psychosocial strengths - prosocial behavior, subjective well-being and impairment in peer relationships, family relationships, and academic/school functioning
2. Exploration of mediation: When comparing SMART and ordinary treatment (TAU), (i) therapeutic alliance is higher in SMART, and (ii) a better treatment effect in SMART is partially mediated by therapeutic alliance

3. Exploration of treatment effect heterogeneity (moderators): Effects of SMART treatment compared to TAU vary between: patients with low versus high level of self-regulation difficulties (full vs partial Developmental trauma disorder), patients with extensive vs less extensive developmental trauma exposure, adolescents (13-17 years) vs younger children (7-12 years), and patients exposed to trauma early in life vs in their teens

At each site, eligible participants are randomized to SMART or ordinary treatment/ TAU. Investigators acquire study data at baseline and outcome data at follow up after 6 and 12 months, and measure therapeutic alliance twice during the treatment process.

DETAILED DESCRIPTION:
Specialized mental health services often fall short in adequate treatment of youth with developmental trauma histories. These youth are often difficult to treat due to composite mental and somatic problems. A promising treatment model for the group is the SMART approach, which utilizes sensory motor therapeutic equipment in a specialized room to support youths' natural ways of regulating bodies and emotions. This may facilitate therapeutic bond, improve regulation of arousal, and facilitate a more effective processing of trauma. The study will test the effectiveness of SMART treatment for young people 7-17 years old with developmental trauma and self-regulation difficulties in a two-group RCT. The investigators hypothesize that the SMART approach is more effective than ordinary treatment for an array of outcome measures, including regulatory capacities, attention and behavior; trauma symptoms; and internalizing and externalizing symptoms. The study also will explore if therapeutic alliance mediates treatment effects and heterogeneity of treatment effects (moderator analyses). The study will include 120 children/ adolescents with developmental trauma exposure and difficulties in self-regulatory capacities from four units at dpt. of child and adolescent mental health, Vestre Viken, randomized to SMART or ordinary treatment. This first RCT of SMART for youth has the potential to test whether the model should be adopted as standard treatment for youth in the target group in Norway and internationally.

ELIGIBILITY:
Inclusion criteria:

These are based on the Developmental Trauma Disorder Semistructured Interview (DTD-SI), which has four domains (A-D). Based on the DTD-SI, which is detailed below, inclusion requires:

* The presence of developmental trauma history (domain A)
* One symptom in each of the domains B-D
* At least four symptoms (of a maximum 15) in domains B-D considered together

Domains A to D above refers to the following:

* Domain A. Lifetime contemporaneous exposure to developmental trauma, defined as either (i) Interpersonal victimization: physical or sexual abuse or assault, domestic/intimate partner violence, bullying, harassment, exploitation, trafficking, hate crimes, or racial/ethnic/identity trauma, or (ii) Primary caregiving system attachment disruption: caregiver change or prolonged separation, gross neglect (physical, medical, emotional), psychological maltreatment (emotional abuse, emotional neglect, parental hostility or over-controlling), caregiver impairment due to mental illness or substance abuse, or chronic medical condition (by child or caregiver)
* Domain B. Affective and somatic dysregulation: (i) Emotion dysregulation, (ii) Somatic dysregulation, (iii) Impaired awareness or dissociation of emotions and body, (iv) Impaired capacity to describe emotions or bodily states
* Domain C. Attentional and behavioral dysregulation: (i) Threat-related rumination, (ii) Impaired capacity for self protection, (iii) Maladaptive self-soothing, (iv) Habitual or reactive self-harm, (v) Inability to initiate or sustain goal-directed behavior
* Domain D. Self and relational dysregulation: (i) Persistent extreme negative self-perception, (ii) attachment insecurity and disorganization, (iii) Extreme persistent distrust, defiance or lack of reciprocity in close relationships, (iv) Reactive physical or verbal aggression, (v) Psychological boundary deficits, (vi) Impaired capacity to regulate empathic arousal

Exclusion Criteria:

* Active psychosis
* Not fluent in Norwegian language
* Developmental challenges - IQ < 70
* Has previously used SMART room

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-regulation difficulties | The outcome is assessed by trained study personell at Baseline (Day 1) and at follow up 6 months and 12 months after Baseline.
  Domains B, C and D on the Developmental trauma disorder semistructured interview (DTD-SI). Scores on DTD-SI range from 0-15, where higher scores mean more self-regulation difficulties (and worse outcome).

SECONDARY OUTCOMES:
International Trauma Questionnaire (ITQ) | The outcome is assessed by trained study personell at Baseline (Day 1) and at follow up 6 months and 12 months after Baseline.
  Core features of PTSD and complex PTSD. We use total scores and subdomain scores. Total scores range from 0-72, where higher scores mean worse outcome. Subdomain scores for each of PTSD and complex PTSD range from 0-36, and also here higher scores mean worse outcome.
Strenght and Difficulties Questionnaire (SDQ) | Assessed at baseline and 6 and 12 months follow up
  Psychosocial problems and strengths, based on assessing five domains: emotional symptoms, conduct problems, hyperactivity-inattention, peer problems, and prosocial behavior. The study will use a total difficulties score based on the first 4 of the 5 subdomains of SDQ, with scores ranging from 0-40, where higher scores mean worse outcome. The study also will use a total score for the fifth domain alone, about psychosocial strenghts, with scores ranging from 0-10 and higher scores meaning better outcome.
Child Behavior Checklist (CBCL/6-18)/ Youth self-report (YRS) from ASEBA | Assessed at baseline and at 6 and 12 months follow up
  CBCL/6-18 / YRS 6-18 consist of 113 behavioral items, scored on a 3-point scale ranging from 0 ("not true") to 2 ("very true" (2). Based on factor analysis and norm data, raw scores are translated into T-scores (0-100, mean 50) for an array of scales by using ASEBA software. The study will use T-scores (or eventually raw scores) for the following scales: (i) Eight syndrome scales (anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, and aggressive behavior); (ii) Total problems - sum of scores from all eight syndrome scales (iii); Externalizing problems (sum of rule-breaking and aggressive behavior scores); (iv) Internalizing problems (sum of anxious/depressed, withdrawn/depressed, and somatic complaints scores), (v); Dysregulation (based on 18 items); (vi) six DSM-IV-oriented scales, and (vii) Adaptive functioning scale (14 items). Higher scores generally mean worse outcome, but opposite for (vii).
Child outcome rating scale (CORS) | Assessed at baseline and at 6 and 12 months follow up
  CORS provides a measure of subjective well-being. CORS consists of 4 items that are scored on a visual analogue scale, with scores for each item ranging from 0-10. Total score on CORS range from 0-40, where higher scores mean better outcome.

OTHER OUTCOMES:
Therapeutic alliance scale for children - revised (TASC-R) | Measured after the 3rd and the 7th psychotherapy treatment session, that is, 3 and 7 weeks after Baseline - since participants will receive one psychotherapy treatment session per week.
  TASC-R is a measure of therapeutic alliance or working alliance. Scores on TASC-R range from 12 to 48, where higher scores mean better outcome
Session rating scale for children (CSRS) | Measured after the 3rd and the 7th psychotherapy treatment session, that is, 3 and 7 weeks after Baseline - since participants will receive one psychotherapy treatment session per week.
  CSRS is a measure of therapeutic alliance or working alliance. Four items are scored on visual analogue scales, each representing scores from 0-10, with total scores on CSRS ranging from 0-40. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Roar Fosse, Ph.D., Principal Investigator — Vestre Viken Hospital Trust
Locations (4):
- Norway (4):
  - Dpt of Child and Adolescent Mental Health (CAMH) Vestre Viken - Asker, Asker, Akershus
  - Dpt of Child and Adolescent Mental Health (CAMH) Vestre Viken - Ringerike Ål, Ål, Buskerud
  - Dpt of Child and Adolescent Mental Health (CAMH) Vestre Viken - Drammen, Drammen, Buskerud
  - Dpt of Child and Adolescent Mental Health (CAMH) Vestre Viken - Kongsberg, Kongsberg, Buskerud

IPD SHARING:
Plan to Share IPD: No